CLINICAL TRIAL: NCT00512928
Title: Safety Study of Vitamin K2 During Anticoagulation in Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Dr. C. Vermeer, VitaK BV
Organization: Maastricht University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 07-3-032
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: vitamin K2; oral anticoagulation; interference; level of anticoagulation; carboxylation level of osteocalcin and matrix-gla protein
MeSH Terms: interventions — Acenocoumarol; menaquinone 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acenocoumarol — max 5 mg per day during 10 weeks
  Other Names: sintrom mitis
Dietary Supplement: menaquinone-7 — In successive weeks (6 weeks) the dosage is increased over the range 10 µg to 20 µg increasing to 45 µg MK-7 for the final week.
  Other Names: MenaQ7

SUMMARY:
Oral anticoagulants that are widely used for the treatment of thrombo-embolic disease exert their effect by blocking the recycling of vitamin K. Vitamin K acts as a co-factor in the posttranslational carboxylation of vitamin K-dependent proteins such as osteocalcin and matrix-gla protein. It is important to quantify the dose-response relationship of the interaction between vitamin K and oral anticoagulants and to investigate at what dosage vitamin K will interfere with oral anticoagulants in a clinically relevant way.

DETAILED DESCRIPTION:
From all K-vitamins, menaquinone-7 has been identified as the most effective cofactor for the carboxylation reaction of Gla-proteins. In this respect it is important to quantify the dose-response relationship of the interaction between oral anticoagulants and menaquinone-7. The primary objective of the study is to demonstrate at what menaquinone-7 intake the vitamin will interfere with oral anticoagulants in a clinically relevant way. Clinically relevant is defined as a decrease in level of anticoagulation that would require a change in oral anticoagulant treatment in order to stay within target levels. Secondary objective of the study is to investigate changes in carboxylation level of osteocalcin and matrix-gla protein after menaquinone-7 supplementation during the oral anticoagulation treatment period. This will demonstrate whether during oral anticoagulation menaquinone-7 will be transported preferentially to the liver or to other target tissues.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between 18 and 45 years of age.
* Subjects of normal body weight and height according to BMI < 30
* Subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with (a history of) of coagulation disorders
* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects using (multi)-vitamin supplements containing vitamin K
* Subjects presenting chronic inflammatory diseases
* Subjects using any medication 3 months prior to the study (e.g. corticoϊd treatment, oral anticoagulants)
* Subjects using oral anticonception
* Subject with (a history of) soy allergy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
changes in level anticoagulation | 10 weeks

SECONDARY OUTCOMES:
changes in carboxylation level of osteocalcin and matrix-gla protein | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands